CLINICAL TRIAL: NCT04212091
Title: A Phase 1 Dose-escalation Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of the Monoclonal Antibody PGT121.414.LS Administered Alone and in Combination With VRC07-523LS Via Intravenous or Subcutaneous Infusions in Healthy, HIV-uninfected Adult Participants
Brief Title: Evaluating the Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of the Monoclonal Antibody PGT121.414.LS Administered Alone and in Combination With VRC07-523LS Via Intravenous or Subcutaneous Infusions in Healthy, HIV-uninfected Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: HIV Vaccine Trials Network (Network); HIV Prevention Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 136/HPTN 092; 38634 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2019-12-23; First posted 2019-12-26 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-05

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A (Group 1): PGT121.414.LS (3 mg/kg) (Experimental): Participants will receive 3 mg/kg of PGT121.414.LS by intravenous (IV) infusion at Month 0.
  Interventions: Biological: PGT121.414.LS
- Part A (Group 2): PGT121.414.LS (10 mg/kg) (Experimental): Participants will receive 10 mg/kg of PGT121.414.LS by IV infusion at Month 0.
  Interventions: Biological: PGT121.414.LS
- Part A (Group 3): PGT121.414.LS (30 mg/kg) (Experimental): Participants will receive 30 mg/kg of PGT121.414.LS by IV infusion at Month 0.
  Interventions: Biological: PGT121.414.LS
- Part A (Group 4): PGT121.414.LS (5 mg/kg) (Experimental): Participants will receive 5 mg/kg of PGT121.414.LS by subcutaneous (SC) infusion at Month 0.
  Interventions: Biological: PGT121.414.LS
- Part B (Group 5): PGT121.414.LS + VRC07-523LS (20 mg/kg) (Experimental): Participants will receive 20 mg/kg of PGT121.414.LS and 20 mg/kg of VRC07-523LS by IV infusion sequentially in this order at Months 0, 4, and 8.
  Interventions: Biological: PGT121.414.LS; Biological: VRC07-523LS
- Part B (Group 6): PGT121.414.LS + VRC07-523LS (5 mg/kg) (Experimental): Participants will receive 5 mg/kg of PGT121.414.LS and 5 mg/kg of VRC07-523LS by SC infusion sequentially in this order at Months 0, 4, and 8.
  Interventions: Biological: PGT121.414.LS; Biological: VRC07-523LS

INTERVENTIONS:
Biological: PGT121.414.LS — Administered via IV infusion or SC infusion, depending on the arm
Biological: VRC07-523LS — Administered via IV infusion or SC infusion, depending on the arm
  Arms: Part B (Group 5): PGT121.414.LS + VRC07-523LS (20 mg/kg); Part B (Group 6): PGT121.414.LS + VRC07-523LS (5 mg/kg)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and antiviral activity of the monoclonal antibody PGT121.414.LS administered alone and in combination with VRC07-523LS via intravenous or subcutaneous infusions in healthy, HIV-uninfected adult participants.

DETAILED DESCRIPTION:
This study will evaluate the safety, tolerability, pharmacokinetics, and antiviral activity of the monoclonal antibody PGT121.414.LS administered alone and in combination with VRC07-523LS via intravenous (IV) or subcutaneous (SC) infusions in healthy, HIV-uninfected adult participants.

The study will be conducted in two parts (Part A and B). Part A will include four groups (Groups 1, 2, 3, and 4) and Part B will include two groups (Groups 5 and 6).

In Part A of the study, PGT121.414.LS will be administered via IV infusion at 3, 10, or 30 mg/kg (Groups 1-3) or via SC infusion at 5 mg/kg (Group 4). Participants in Part B will receive consecutive administration of PGT121.414.LS followed by VRC07-523LS, at 20 mg/kg IV each per dose (Group 5) or 5 mg/kg SC each per dose (Group 6). Participants will be followed for 32 weeks after the last study product administration via IV infusion and 24 weeks after the last study product administration via SC infusion.

Participants in Groups 1, 2, and 3 will attend 8 months of study visits. Participants in Group 4 will attend 6 months of study visits. Part B participants will attend 16 months of study visits. Study visits may include physical examinations, blood and urine collection, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria

* Age of 18 to 50 years
* Access to a participating Clinical Research Site (CRS) and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Assessment of understanding: volunteer demonstrates understanding of this study and completes a questionnaire prior to first study product administration with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Agrees not to enroll in another study of an investigational research agent until completion of the last required protocol clinic visit
* Good general health as shown by medical history, physical exam, and screening laboratory tests

HIV-Related Criteria:

* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling.
* Assessed by the clinic staff as being at "low risk" for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit (see study protocol).

Laboratory Inclusion Values:

Hemogram/Complete Blood Count

* Hemoglobin ≥11.0 g/dL for participants who were assigned female sex at birth, ≥13.0 g/dL for participants who were assigned male sex at birth. For transgender participants who have been on feminizing hormone therapy for more than 6 consecutive months, determine hemoglobin eligibility based on the gender with which they identify (ie, a transgender female who has been on hormone therapy for more than 6 consecutive months should be assessed for eligibility using the hemoglobin parameters for persons assigned female sex at birth).
* White blood cell (WBC) count = 2,500 to 12,000 cells/mm^3
* WBC differential either within institutional normal range or with site clinician approval
* Platelets = 125,000 to 550,000 cells/mm^3

Chemistry

* Chemistry panel: alanine aminotransferase (ALT) <1.25 times the institutional upper limit of normal; creatinine ≤ institutional upper limit of normal

Virology

* Negative HIV-1 and -2 blood test: US volunteers must have a negative Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA) or chemiluminescent microparticle immunoassay (CMIA).
* Negative Hepatitis B surface antigen (HBsAg)
* Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive

Urine

* Negative or trace urine protein

Reproductive Status

* Volunteers who were assigned female sex at birth: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test performed prior to study product administration on the day of initial study product administration. Persons who are NOT of reproductive potential due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing
* Reproductive status: A volunteer who was assigned female sex at birth must:

  * Agree to use effective contraception for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit. Effective contraception is defined as using the following methods:
  * Condoms (male or female) with or without a spermicide,
  * Diaphragm or cervical cap with spermicide,
  * Intrauterine device (IUD),
  * Hormonal contraception,
  * Tubal ligation, or
  * Any other contraceptive method approved by the HIV Vaccine Trials Network (HVTN) 136/HIV Prevention Trials Network (HPTN) 092 Protocol Safety Review Team (PSRT)
  * Successful vasectomy in any partner assigned male sex at birth (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy);
  * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy;
  * Or be sexually abstinent.
* Volunteers who were assigned female sex at birth must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Exclusion Criteria:

General

* Weight >115 kg
* Blood products received within 120 days before first study product administration, unless eligibility for earlier enrollment is determined by the HVTN 136/HPTN 092 PSRT
* Investigational research agents received within 30 days before first study product administration
* Intent to participate in another study of an investigational research agent or any other study that requires non-Network HIV antibody testing during the planned duration of the study
* Pregnant or breastfeeding

Vaccines and other Injections

* HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 136/HPTN 092 PSRT will determine eligibility on a case-by-case basis.
* Previous receipt of humanized or human mAbs, whether licensed or investigational; the HVTN 136/HPTN 092 PSRT will determine eligibility on a case-by-case basis.
* Previous receipt of monoclonal antibodies VRC01, VRC01LS, VRC07-523LS, or PGT121

Immune System

* Immunosuppressive medications received within 30 days before first study product administration (Not exclusionary: [1] corticosteroid nasal spray; [2] inhaled corticosteroids; [3] topical corticosteroids for mild, uncomplicated dermatological condition; or [4] a single course of oral/parenteral prednisone or equivalent at doses <20 mg/day and length of therapy <14 days.)
* Serious adverse reactions to VRC07-523LS or PGT121.414.LS formulation components (acetate, sucrose, polysorbate 80, histidine, and sorbitol; see study protocol), including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain
* Immunoglobulin received within 90 days before first study product administration, unless eligibility for earlier enrollment is determined by the HVTN 136/HPTN 092 PSRT (for mAb see criterion above)
* Autoimmune disease (Not excluded from participation: Participant with mild, stable and uncomplicated autoimmune disease that does not require immunosuppressive medication and that, in the judgment of the site investigator, is likely not subject to exacerbation and likely not to complicate Solicited and Unsolicited AE assessments)
* Immunodeficiency

Clinically significant medical conditions

* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response,
  * A process that would require medication that affects the immune response,
  * Any contraindication to repeated infusions, or blood draws, including inability to establish venous or subcutaneous access,
  * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
  * A condition or process (eg, chronic urticaria or recent injection or infusion with evidence of residual inflammation) for which signs or symptoms could be confused with reactions to the study product, or
  * Any condition specifically listed among the exclusion criteria.
* Any medical, psychiatric, occupational, or skin condition (eg, tattoos) that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety, Solicited AEs, or a participant's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis (TB) therapy
* Asthma other than mild, well-controlled asthma. (Symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program (NAEPP) Expert Panel report).
* Exclude a volunteer who:

  * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
  * Uses moderate/high-dose, inhaled corticosteroids, or
* In the past year has either of the following:

  * Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids;
  * Needed emergency care, urgent care, hospitalization, or intubation for asthma.
* Diabetes mellitus type 1 or type 2 (Not excluded: type 2 cases controlled with diet alone or a history of isolated gestational diabetes.)
* Hypertension:

  * If a person has been found to have elevated blood pressure or hypertension during screening or previously, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently ≤140 mm Hg systolic and ≤90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be ≤150 mm Hg systolic and ≤100 mm Hg diastolic. For these volunteers, blood pressure must be ≤140 mm Hg systolic and ≤90 mm Hg diastolic at enrollment.
  * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure ≥150 mm Hg at enrollment or diastolic blood pressure ≥100 mm Hg at enrollment.
* Bleeding disorder diagnosed by a clinician (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (Not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study)
* Seizure disorder: History of seizure(s) within past 3 years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Asplenia: any condition resulting in the absence of a functional spleen
* History of generalized urticaria, angioedema, or anaphylaxis.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hurt, Study Chair — University of North Carolina, Chapel Hill; Kathryn Stephenson, Study Chair — Beth Israel Deaconess Medical Center, Harvard University; Srilatha Edupuganti, Study Chair — Emory University
Locations (5):
- United States (5):
  - UCLA CARE Center CRS, Los Angeles, California
  - George Washington Univ. CRS, Washington D.C., District of Columbia
  - The Hope Clinic of the Emory Vaccine Center CRS, Decatur, Georgia
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Columbia P&S CRS, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Edupuganti S, Hurt CB, Stephenson KE, Huang Y, Paez CA, Yu C, Yen C, Hanscom B, He Z, Miner MD, Gamble T, Heptinstall J, Seaton KE, Domin E, Lin BC, McKee K, Doria-Rose N, Regenold S, Spiegel H, Anderson M, McClosky N, Zhang L, Piwowar-Manning E, Ackerman ME, Pensiero M, Dye BJ, Landovitz RJ, Mayer K, Siegel M, Sobieszczyk M, Walsh SR, Gama L, Barouch DH, Montefiori DC, Tomaras GD; HVTN 136/HPTN 092 Study Team. Safety, tolerability, pharmacokinetics, and neutralisation activities of the anti-HIV-1 monoclonal antibody PGT121.414.LS administered alone and in combination with VRC07-523LS in adults without HIV in the USA (HVTN 136/HPTN 092): a first-in-human, open-label, randomised controlled phase 1 trial. Lancet HIV. 2025 Jan;12(1):e13-e25. doi: 10.1016/S2352-3018(24)00247-9. Epub 2024 Dec 10. PMID 39667379

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant enrolled in Group 2 was later deemed ineligible due to a preexisting autoimmune condition that required immunosuppressive treatment at the time of enrollment. The participant was included in the PK, neutralization, and ADA analysis but was excluded from the safety analysis.
Groups:
- Group 1: Vaccine: PGT121.414.LS 3 mg/kg IV mo(0)
- Group 2: Vaccine: PGT121.414.LS 10 mg/kg IV mo(0)
- Group 3: Vaccine: PGT121.414.LS 30 mg/kg IV mo(0)
- Group 4: Vaccine: PGT121.414.LS 5 mg/kg SC mo(0)
- Group 5: Vaccine: PGT121.414.LS 20 mg/kg and VRC07-523LS 20 mg/kg IV sequentially at Mo(0, 4, 8)
- Group 6: Vaccine: PGT121.414.LS 5 mg/kg and VRC07-523LS 5 mg/kg SC sequentially at Mo(0, 4, 8)
Period: Overall Study
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine
Started | 3 | 4 | 3 | 3 | 10 | 10
Completed | 3 | 4 | 3 | 3 | 8 | 9
Not Completed | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Participant unable to adhere to visit | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine | Total
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 10 | 10 | 33
Age, Continuous [Median (Full Range); unit: years] | 29 [22 to 37] | 29 [24 to 31] | 39 [30 to 40] | 39 [25 to 48] | 34 [24 to 41] | 29 [24 to 43] | 31 [22 to 48]
Age, Customized [Count of Participants; unit: Participants]
  Less than 18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18 - 20 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  21 - 30 years | 2 | 2 | 1 | 1 | 3 | 5 | 14
  31 - 40 years | 1 | 2 | 2 | 1 | 6 | 4 | 16
  41 - 50 years | 0 | 0 | 0 | 1 | 1 | 1 | 3
  Above 50 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 2 | 2 | 6 | 3 | 19
  Male | 1 | 0 | 1 | 1 | 4 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 3 | 1 | 4
  Not Hispanic or Latino | 3 | 4 | 3 | 3 | 7 | 9 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 1 | 0 | 0 | 1 | 0 | 0 | 2
  White | 2 | 4 | 3 | 2 | 9 | 7 | 27
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  USA | 3 | 4 | 3 | 3 | 10 | 10 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Pain and/or Tenderness
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [July 2017]. The maximum grade observed for each symptom over the time frame is presented
Time Frame: Measured through 3 days after each vaccine dose at T1-T4: Day 0; T5-T6: Days 0, 112, 224
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 10 | 10
Participants
  None | 3 | 3 | 3 | 3 | 4 | 3
  Mild | 0 | 0 | 0 | 0 | 4 | 7
  Moderate | 0 | 0 | 0 | 0 | 2 | 0
  Severe | 0 | 0 | 0 | 0 | 0 | 0
  Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms: Erythema and/or Induration
Description: as for outcome 1
Time Frame: Measured through 3 days after each vaccine dose at T1-T4: Day 0; T5-T6: Days 0, 112, 224
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 10 | 10
Participants
  Erythema/Redness: None | 3 | 3 | 3 | 3 | 10 | 4
  Erythema/Redness: Mild | 0 | 0 | 0 | 0 | 0 | 4
  Erythema/Redness: Moderate | 0 | 0 | 0 | 0 | 0 | 2
  Erythema/Redness: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Erythema/Redness: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Induration/Swelling: None | 3 | 3 | 3 | 3 | 10 | 4
  Induration/Swelling: Mild | 0 | 0 | 0 | 0 | 0 | 4
  Induration/Swelling: Moderate | 0 | 0 | 0 | 0 | 0 | 2
  Induration/Swelling: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Induration/Swelling: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Erythema and/or Induration: None | 3 | 3 | 3 | 3 | 10 | 4
  Erythema and/or Induration: Mild | 0 | 0 | 0 | 0 | 0 | 4
  Erythema and/or Induration: Moderate | 0 | 0 | 0 | 0 | 0 | 2
  Erythema and/or Induration: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Erythema and/or Induration: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1 [July 2017]. The following symptoms are considered as systemic reactogenicity if the onset date was within the periods of assessment specified in the protocol: malaise and/or fatigue, myalgia, headache, nausea, vomiting, chills, arthralgia, and body temperature. The item Max. Systemic Symptoms is the maximum of the individual systemic reactogenicities excluding body temperature for a participant
Time Frame: Measured through 3 days after each vaccine dose at T1-T4: Day 0; T5-T6: Days 0, 112, 224
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 10 | 10
Participants
  Malaise and/or fatigue: None | 3 | 1 | 2 | 2 | 4 | 5
  Malaise and/or fatigue: Mild | 0 | 2 | 1 | 1 | 4 | 4
  Malaise and/or fatigue: Moderate | 0 | 0 | 0 | 0 | 2 | 1
  Malaise and/or fatigue: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Malaise and/or fatigue: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: None | 3 | 3 | 3 | 2 | 8 | 9
  Myalgia: Mild | 0 | 0 | 0 | 1 | 2 | 1
  Myalgia: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Myalgia: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Headache: None | 3 | 2 | 1 | 3 | 3 | 8
  Headache: Mild | 0 | 1 | 2 | 0 | 5 | 2
  Headache: Moderate | 0 | 0 | 0 | 0 | 2 | 0
  Headache: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Headache: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: None | 2 | 3 | 3 | 3 | 7 | 9
  Nausea: Mild | 1 | 0 | 0 | 0 | 3 | 1
  Nausea: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Nausea: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Chills: None | 3 | 3 | 3 | 3 | 8 | 10
  Chills: Mild | 0 | 0 | 0 | 0 | 2 | 0
  Chills: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Chills: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Chills: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: None | 3 | 3 | 3 | 3 | 8 | 10
  Arthralgia: Mild | 0 | 0 | 0 | 0 | 2 | 0
  Arthralgia: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Arthralgia: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Urticaria: None | 3 | 3 | 3 | 3 | 10 | 10
  Urticaria: Mild | 0 | 0 | 0 | 0 | 0 | 0
  Urticaria: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Urticaria: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Urticaria: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Generalized Pruritus: None | 3 | 3 | 3 | 3 | 10 | 10
  Generalized Pruritus: Mild | 0 | 0 | 0 | 0 | 0 | 0
  Generalized Pruritus: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Generalized Pruritus: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Generalized Pruritus: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Max. Systemic Symptoms: None | 2 | 1 | 1 | 2 | 2 | 5
  Max. Systemic Symptoms: Mild | 1 | 2 | 2 | 1 | 5 | 4
  Max. Systemic Symptoms: Moderate | 0 | 0 | 0 | 0 | 3 | 1
  Max. Systemic Symptoms: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Max. Systemic Symptoms: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: None | 3 | 3 | 3 | 3 | 10 | 9
  Temperature: Mild | 0 | 0 | 0 | 0 | 0 | 1
  Temperature: Moderate | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: Severe | 0 | 0 | 0 | 0 | 0 | 0
  Temperature: Potentially Life-threatening | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Chemistry and Hematology Laboratory Measures - Alkaline Phosphatase, AST, ALT in U/L
Description: For each local laboratory measure, summary statistics were presented by treatment group and timepoint for the overall population
Time Frame: Measured during Screening, Days 0, 112, 168
Population: 'Overall Number of Participants Analyzed' represents participants enrolled and eligible for laboratory assessment. Participants do not have laboratory assessments if they attended the visit but laboratory specimens were not collected, missed the scheduled visit, or terminated participation in the study prior to the scheduled visit. AST and Alkaline Phosphatase data were not collected at screening.
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 10 | 10
U/L
  ALT (SGPT) (U/L)- Screening | 14.0 [11.0 to 23.0] | 14.0 [12.0 to 18.0] | 14.0 [14.0 to 24.0] | 17.0 [12.0 to 19.0] | 13.0 [12.0 to 18.0] | 16.0 [11.0 to 24.0]
  ALT (SGPT) (U/L)- Day 0/Enrollment | 17.0 [11.0 to 25.0] | 13.0 [12.0 to 16.0] | 15.0 [14.0 to 23.0] | 14.0 [13.0 to 17.0] | 15.0 [13.0 to 23.0] | 15.5 [12.0 to 22.0]
  ALT (SGPT) (U/L)- Day 112: number analyzed (Participants) | 3 | 3 | 3 | 3 | 9 | 10
  ALT (SGPT) (U/L)- Day 112 | 13.0 [10.0 to 21.0] | 15.0 [10.0 to 19.0] | 14.0 [13.0 to 21.0] | 15.0 [12.0 to 19.0] | 15.0 [13.0 to 18.0] | 18.0 [9.0 to 26.0]
  ALT (SGPT) (U/L)- Day 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 10 | 9
  ALT (SGPT) (U/L)- Day 168 | 12.0 [12.0 to 20.0] | 17.0 [11.0 to 18.0] | 15.0 [12.0 to 20.0] | 13.0 [13.0 to 21.0] | 20.0 [15.0 to 21.0] | 15.0 [11.0 to 19.0]
  AST (U/L)- Day 0/Enrollment | 18.0 [14.0 to 23.0] | 20.0 [19.0 to 22.0] | 18.0 [16.0 to 19.0] | 19.0 [14.0 to 20.0] | 19.0 [16.0 to 23.0] | 17.0 [13.0 to 24.0]
  AST (U/L)- Day 112: number analyzed (Participants) | 3 | 3 | 3 | 3 | 9 | 10
  AST (U/L)- Day 112 | 16.0 [15.0 to 19.0] | 21.0 [15.0 to 24.0] | 16.0 [13.0 to 22.0] | 15.0 [15.0 to 32.0] | 19.0 [17.0 to 20.0] | 19.0 [15.0 to 24.0]
  AST (U/L)- Day 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 10 | 9
  AST (U/L)- Day 168 | 15.0 [14.0 to 19.0] | 23.0 [19.0 to 23.0] | 15.0 [14.0 to 21.0] | 15.0 [12.0 to 24.0] | 19.0 [18.0 to 21.0] | 17.0 [15.0 to 18.0]
  Alkaline Phosphatase(U/L)- Day 0/Enrollment | 55.0 [52.0 to 77.0] | 46.0 [43.0 to 59.0] | 57.0 [36.0 to 72.0] | 63.0 [40.0 to 72.0] | 61.5 [54.0 to 76.0] | 58.0 [50.0 to 75.0]
  Alkaline Phosphatase(U/L)- Day 112: number analyzed (Participants) | 3 | 3 | 3 | 3 | 9 | 10
  Alkaline Phosphatase(U/L)- Day 112 | 57.0 [55.0 to 77.0] | 52.0 [46.0 to 65.0] | 55.0 [45.0 to 80.0] | 60.0 [38.0 to 72.0] | 68.0 [61.0 to 70.0] | 57.5 [41.0 to 71.0]
  Alkaline Phosphatase(U/L)- Day 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 10 | 9
  Alkaline Phosphatase(U/L)- Day 168 | 57.0 [55.0 to 72.0] | 57.0 [40.0 to 65.0] | 54.0 [37.0 to 79.0] | 57.0 [39.0 to 71.0] | 73.5 [62.0 to 81.0] | 58.0 [50.0 to 79.0]

5. Primary Outcome: Chemistry and Hematology Laboratory Measures - Creatinine in mg/dL
Description: as for outcome 4
Time Frame: Measured during Screening, Days 0, 112, 168
Population: 'Overall Number of Participants Analyzed' represents participants enrolled and eligible for laboratory assessment. Participants do not have laboratory assessments if they attended the visit but laboratory specimens were not collected, missed the scheduled visit, or terminated participation in the study prior to the scheduled visit.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 10 | 10
mg/dL
  Creatinine (g/dL)- Screening | 1.0200 [.86000 to 1.1700] | .60000 [.46000 to .83000] | .97000 [.85000 to 1.0400] | .73000 [.72000 to .87000] | .78500 [.63000 to .86000] | .89000 [.78000 to .95000]
  Creatinine (g/dL)- Day 0/Enrollment | .90000 [.80000 to 1.0800] | .70000 [.58000 to .71000] | .94000 [.78000 to 1.1200] | .75000 [.66000 to .97000] | .78000 [.71000 to .85000] | .82000 [.71000 to 1.0000]
  Creatinine (g/dL)- Day 112: number analyzed (Participants) | 3 | 3 | 3 | 3 | 9 | 10
  Creatinine (g/dL)- Day 112 | .91000 [.68000 to 1.1500] | .68000 [.59000 to .81000] | .94000 [.78000 to 1.3100] | .81000 [.78000 to .99000] | .80000 [.77000 to .88000] | .79000 [.65000 to .97000]
  Creatinine (g/dL)- Day 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 10 | 9
  Creatinine (g/dL)- Day 168 | .81000 [.61000 to 1.0800] | .71000 [.60000 to .82000] | .90000 [.85000 to 1.0300] | .82000 [.68000 to .96000] | .82000 [.70000 to .92000] | .83000 [.79000 to .97000]

6. Primary Outcome: Chemistry and Hematology Laboratory Measures - Hemoglobin in g/dL
Description: as for outcome 4
Time Frame: Measured during Screening, Days 0, 112, 168
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 10 | 10
g/dL
  Hemoglobin (g/dL)- Screening | 14.1 [12.7 to 16.7] | 13.1 [11.1 to 13.7] | 13.8 [13.0 to 16.4] | 12.9 [11.3 to 14.9] | 13.6 [12.1 to 14.7] | 14.1 [13.5 to 14.8]
  Hemoglobin (g/dL)- Day 0/Enrollment | 13.5 [11.4 to 17.7] | 12.9 [11.2 to 13.2] | 13.4 [12.4 to 16.7] | 12.4 [11.5 to 15.0] | 12.6 [12.1 to 14.6] | 14.2 [13.0 to 15.0]
  Hemoglobin (g/dL)- Day 112: number analyzed (Participants) | 3 | 3 | 3 | 3 | 9 | 10
  Hemoglobin (g/dL)- Day 112 | 13.9 [12.5 to 16.6] | 12.9 [12.4 to 13.7] | 14.2 [12.5 to 14.4] | 12.7 [10.1 to 14.1] | 12.6 [11.5 to 14.7] | 14.1 [12.9 to 15.4]
  Hemoglobin (g/dL)- Day 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 10 | 9
  Hemoglobin (g/dL)- Day 168 | 13.5 [12.1 to 17.3] | 13.3 [12.2 to 13.5] | 14.0 [11.8 to 14.8] | 12.3 [10.9 to 14.4] | 12.7 [12.4 to 14.3] | 14.2 [13.5 to 14.6]

7. Primary Outcome: Chemistry and Hematology Laboratory Measures - Lymphocyte Count, Neutrophil Count in 1000 Cells/Cubic mm
Description: as for outcome 4
Time Frame: Measured during Screening, Days 0, 112, 168
Population: "Overall Number of Participants Analyzed" represents participants enrolled and eligible for laboratory assessment. Participants do not have laboratory assessments if they attended the visit but laboratory specimens were not collected, missed the scheduled visit, or terminated participation in the study prior to the scheduled visit.
Measure: Median (Inter-Quartile Range); unit: 1000 cells/cubic mm
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 10 | 10
1000 cells/cubic mm
  Neutrophils (1000 cells/cubic mm)- Screening | 5.05 [1.80 to 9.42] | 4.31 [3.80 to 4.92] | 2.83 [2.07 to 4.90] | 4.20 [2.05 to 7.33] | 3.92 [2.80 to 5.39] | 3.50 [2.37 to 5.12]
  Neutrophils (1000 cells/cubic mm)- Day 0/Enrollment | 2.60 [1.70 to 3.95] | 3.59 [3.29 to 5.80] | 2.88 [1.63 to 4.20] | 3.70 [2.40 to 6.09] | 4.01 [2.53 to 4.36] | 3.32 [2.22 to 4.52]
  Neutrophils (1000 cells/cubic mm)- Day 112: number analyzed (Participants) | 3 | 3 | 3 | 3 | 9 | 10
  Neutrophils (1000 cells/cubic mm)- Day 112 | 3.80 [1.90 to 5.06] | 4.20 [2.66 to 4.38] | 2.11 [1.84 to 3.80] | 3.50 [1.99 to 5.26] | 3.65 [2.59 to 5.77] | 3.26 [3.06 to 5.32]
  Neutrophils (1000 cells/cubic mm)- Day 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 10 | 9
  Neutrophils (1000 cells/cubic mm)- Day 168 | 4.51 [2.50 to 5.93] | 4.37 [4.04 to 5.20] | 2.42 [1.88 to 4.90] | 3.20 [2.01 to 5.72] | 3.71 [3.17 to 4.50] | 2.88 [2.59 to 4.39]
  Lymphocytes (1000 cells/cubic mm)- Screening | 2.14 [1.17 to 2.20] | 2.06 [1.86 to 2.30] | 2.10 [1.23 to 4.15] | 2.00 [1.66 to 2.70] | 2.06 [1.70 to 2.30] | 1.68 [1.24 to 1.91]
  Lymphocytes (1000 cells/cubic mm)- Day 0/Enrollment | 2.26 [2.22 to 2.60] | 1.55 [1.46 to 2.20] | 1.90 [1.44 to 3.04] | 1.98 [1.68 to 2.00] | 1.68 [1.40 to 2.28] | 1.89 [1.33 to 2.30]
  Lymphocytes (1000 cells/cubic mm)- Day 112: number analyzed (Participants) | 3 | 3 | 3 | 3 | 9 | 10
  Lymphocytes (1000 cells/cubic mm)- Day 112 | 2.20 [1.72 to 2.40] | 1.66 [1.31 to 2.80] | 2.12 [1.96 to 2.20] | 1.99 [1.46 to 2.10] | 1.76 [1.48 to 2.06] | 1.81 [1.47 to 1.92]
  Lymphocytes (1000 cells/cubic mm)- Day 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 10 | 9
  Lymphocytes (1000 cells/cubic mm)- Day 168 | 2.10 [1.75 to 2.59] | 1.99 [1.89 to 2.70] | 2.40 [1.44 to 2.70] | 1.65 [1.56 to 2.30] | 1.68 [1.55 to 2.24] | 1.86 [1.67 to 2.10]

8. Primary Outcome: Chemistry and Hematology Laboratory Measures - Platelets, WBC in 1000 Cells/Cubic mm
Description: as for outcome 4
Time Frame: Measured during Screening, Days 0, 112, 168
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: 1000 cells/cubic mm
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 10 | 10
1000 cells/cubic mm
  WBC (1000 cells/cubic mm)- Screening | 7.80 [4.50 to 10.90] | 7.20 [6.80 to 7.30] | 7.70 [3.71 to 8.00] | 7.50 [4.33 to 10.30] | 6.37 [5.09 to 8.02] | 5.46 [4.20 to 7.95]
  WBC (1000 cells/cubic mm)- Day 0/Enrollment | 5.60 [4.70 to 6.80] | 5.70 [5.60 to 8.70] | 6.70 [3.51 to 6.90] | 6.20 [4.61 to 9.00] | 6.28 [5.44 to 7.43] | 5.63 [4.69 to 7.27]
  WBC (1000 cells/cubic mm)- Day 112: number analyzed (Participants) | 3 | 3 | 3 | 3 | 9 | 10
  WBC (1000 cells/cubic mm)- Day 112 | 6.60 [4.70 to 7.40] | 6.90 [4.60 to 7.60] | 4.80 [4.59 to 6.90] | 6.40 [4.70 to 7.60] | 5.95 [4.54 to 8.06] | 5.89 [5.10 to 6.82]
  WBC (1000 cells/cubic mm)- Day 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 10 | 9
  WBC (1000 cells/cubic mm)- Day 168 | 6.90 [5.00 to 9.50] | 7.30 [6.50 to 8.70] | 6.10 [3.75 to 8.40] | 6.10 [4.36 to 8.20] | 6.73 [5.12 to 6.95] | 6.38 [4.71 to 9.10]
  Platelets (1000 cells/cubic mm)- Screening | 234 [203 to 281] | 307 [251 to 353] | 252 [250 to 274] | 303 [195 to 372] | 297 [268 to 314] | 253 [234 to 365]
  Platelets (1000 cells/cubic mm)- Day 0/Enrollment | 229 [185 to 254] | 273 [222 to 379] | 244 [241 to 290] | 296 [183 to 297] | 273 [260 to 287] | 271 [259 to 293]
  Platelets (1000 cells/cubic mm)- Day 112: number analyzed (Participants) | 3 | 3 | 3 | 3 | 9 | 10
  Platelets (1000 cells/cubic mm)- Day 112 | 246 [221 to 330] | 271 [240 to 403] | 291 [266 to 294] | 296 [189 to 339] | 290 [249 to 307] | 284 [255 to 323]
  Platelets (1000 cells/cubic mm)- Day 168: number analyzed (Participants) | 3 | 3 | 3 | 3 | 10 | 9
  Platelets (1000 cells/cubic mm)- Day 168 | 226 [187 to 253] | 313 [248 to 380] | 266 [237 to 331] | 296 [178 to 406] | 297 [265 to 317] | 291 [256 to 334]

9. Primary Outcome: Number of Participants Reporting Unsolicited Adverse Events (AEs)
Description: The number (percentage) of Participants Reporting Unsolicited Adverse Events (AEs) was summarized by arm
Time Frame: Measured through Month 24
Population: Max severity reported per participant over visit
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 10 | 10
Participants
  Mild | 2 | 2 | 1 | 2 | 2 | 0
  Moderate | 1 | 0 | 1 | 0 | 6 | 8
  Severe | 0 | 0 | 0 | 0 | 0 | 0
  Potentially life-threatening | 0 | 0 | 0 | 0 | 0 | 0
  No AE reported | 0 | 1 | 1 | 1 | 2 | 2

10. Primary Outcome: Number of Participants With Early Discontinuation of Vaccinations and Reason for Discontinuation
Description: The number (percentage) of participants with early discontinuation of vaccinations and reason for discontinuation was summarized by arm
Time Frame: Measured through Month 8
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 10 | 10
Participants
  Participant unable to adhere to visit schedule | 0 | 0 | 0 | 0 | 0 | 1
  Unsolicited adverse event | 0 | 0 | 0 | 0 | 3 | 0
  PSRT decision | 0 | 0 | 0 | 0 | 0 | 1
  Did not discontinue SPA | 3 | 3 | 3 | 3 | 7 | 8

11. Primary Outcome: Number of Participants With Early Study Termination and Reason for Early Study Termination
Description: The number (percentage) of participants with early study termination and reason for early study termination was summarized by arm
Time Frame: Measured through Month 16
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 10 | 10
Participants
  Participant unable to adhere to visit schedule | 0 | 0 | 0 | 0 | 1 | 0
  Unable to contact participant | 0 | 0 | 0 | 0 | 1 | 1
  Scheduled exit visit/end of study | 3 | 3 | 3 | 3 | 8 | 9

12. Primary Outcome: PGT121.414.LS and VRC07523LS Serum Concentrations
Description: Serum concentrations of PGT121.414.LS and VRC07-523LS at prespecified timepoints among participants who received all scheduled product administrations
Time Frame: Days 0, 0.0417, 1, 2, 3, 6, 14, 28, 56, 84, 112, 112.0417, 140, 168, 196, 224, 224.0417, 252, 280, 336, 392, 448
Population: Overall Number of Participants Analyzed represents the number of enrolled participants. Number Analyzed shows the number of participants with available data after filtering for assay specific quality control criteria at each timepoint.
Measure: Median (Inter-Quartile Range); unit: ug/ml
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 10 | 10
ug/ml
  PGT121.414.LS-D0 | 0.32666 [0.212155 to 0.408441] | 0.09765 [0.09765 to 0.09765] | 0.09765 [0.09765 to 0.09765] | 0.09765 [0.09765 to 0.09765] | 0.09765 [0.09765 to 0.09765] | 0.09765 [0.09765 to 0.09765]
  PGT121.414.LS-D0.0417: number analyzed (Participants) | 3 | 4 | 3 | 3 | 10 | 8
  PGT121.414.LS-D0.0417 | 63.83584 [63.05451 to 69.88950] | 221.7834 [213.0117 to 240.7665] | 554.8116 [521.6919 to 676.4573] | 0.09765 [0.09765 to 0.206709] | 714.2483 [675.8913 to 842.2093] | 0.868341 [0.501508 to 1.069614]
  PGT121.414.LS-D1: number analyzed (Participants) | 3 | 4 | 3 | 3 | 8 | 0
  PGT121.414.LS-D1 | 57.19892 [53.42500 to 64.15473] | 164.7475 [152.5291 to 186.0908] | 525.8889 [490.3319 to 624.0825] | 15.57179 [10.89182 to 17.40282] | 540.5799 [493.9560 to 597.8813] |
  PGT121.414.LS-D112: number analyzed (Participants) | 3 | 4 | 3 | 3 | 9 | 10
  PGT121.414.LS-D112 | 12.18623 [11.62024 to 12.73220] | 31.38540 [28.27068 to 36.24888] | 113.6597 [96.48752 to 120.9419] | 10.28579 [9.944198 to 12.06092] | 91.12431 [74.69536 to 104.4369] | 14.53687 [13.39469 to 16.86138]
  PGT121.414.LS-D112.0417: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 10
  PGT121.414.LS-D112.0417 |  |  |  |  | 866.2283 [793.2392 to 922.8176] | 13.15082 [12.43524 to 15.52181]
  PGT121.414.LS-D14 | 33.50825 [30.85342 to 36.28367] | 93.52175 [89.45039 to 98.44224] | 287.3416 [266.9812 to 302.3751] | 27.97899 [22.78709 to 34.31463] | 250.1545 [217.2386 to 279.6561] | 45.60168 [40.84005 to 55.71133]
  PGT121.414.LS-D140: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 9
  PGT121.414.LS-D140 |  |  |  |  | 274.8957 [218.4848 to 327.5700] | 53.56555 [52.04341 to 56.40598]
  PGT121.414.LS-D168: number analyzed (Participants) | 3 | 4 | 3 | 3 | 10 | 9
  PGT121.414.LS-D168 | 6.985977 [6.696763 to 7.061191] | 17.03774 [13.97447 to 21.98945] | 70.64411 [58.95990 to 72.42533] | 6.447051 [6.015901 to 7.8547] | 196.5922 [165.2391 to 242.2765] | 40.64268 [36.83466 to 43.96372]
  PGT121.414.LS-D196: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 10
  PGT121.414.LS-D196 |  |  |  |  | 131.9651 [109.7402 to 155.0229] | 30.01136 [26.97888 to 35.25343]
  PGT121.414.LS-D2: number analyzed (Participants) | 3 | 4 | 3 | 3 | 0 | 0
  PGT121.414.LS-D2 | 47.33316 [46.00456 to 54.73760] | 146.6062 [134.8796 to 160.8884] | 501.1791 [437.2141 to 553.0405] | 19.73051 [15.06059 to 26.21644] |  |
  PGT121.414.LS-D224: number analyzed (Participants) | 3 | 4 | 3 | 0 | 9 | 9
  PGT121.414.LS-D224 | 4.546627 [4.249129 to 4.606805] | 11.50982 [8.860303 to 15.35904] | 51.03267 [39.45568 to 54.68444] |  | 100.3895 [83.59215 to 134.0949] | 20.24181 [18.06964 to 22.66155]
  PGT121.414.LS-D224.0417: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 8
  PGT121.414.LS-D224.0417 |  |  |  |  | 858.8545 [767.1668 to 937.6442] | 19.81756 [14.01395 to 22.69359]
  PGT121.414.LS-D252: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 9
  PGT121.414.LS-D252 |  |  |  |  | 300.5559 [101.1321 to 355.2648] | 49.82065 [47.13868 to 61.15881]
  PGT121.414.LS-D28: number analyzed (Participants) | 3 | 3 | 3 | 3 | 10 | 10
  PGT121.414.LS-D28 | 24.41258 [23.89791 to 27.52718] | 86.60540 [82.86720 to 91.74298] | 250.3132 [240.6387 to 279.1332] | 22.88940 [20.97324 to 26.82628] | 218.4120 [175.2238 to 233.6124] | 38.72047 [36.35462 to 48.21425]
  PGT121.414.LS-D280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 8
  PGT121.414.LS-D280 |  |  |  |  | 190.1484 [106.4923 to 211.1041] | 39.22639 [32.07971 to 49.07706]
  PGT121.414.LS-D3: number analyzed (Participants) | 3 | 4 | 3 | 3 | 7 | 10
  PGT121.414.LS-D3 | 42.63419 [41.91706 to 48.18462] | 135.5188 [120.8723 to 153.3014] | 496.2948 [402.0094 to 543.2997] | 21.51805 [17.73029 to 30.87779] | 328.0125 [290.1827 to 413.4903] | 43.11783 [40.49056 to 56.40417]
  PGT121.414.LS-D336: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 9
  PGT121.414.LS-D336 |  |  |  |  | 122.0257 [82.59510 to 146.5593] | 25.60772 [20.73072 to 28.07847]
  PGT121.414.LS-D392: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 9
  PGT121.414.LS-D392 |  |  |  |  | 69.69947 [43.23930 to 95.21436] | 14.40051 [10.43843 to 15.51276]
  PGT121.414.LS-D448: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 0
  PGT121.414.LS-D448 |  |  |  |  | 53.10780 [31.55871 to 59.34636] |
  PGT121.414.LS-D56 | 20.04609 [19.38634 to 20.85822] | 59.34368 [55.10586 to 63.75242] | 185.9332 [178.5389 to 213.6618] | 19.82906 [16.27034 to 21.76373] | 152.5493 [117.0020 to 162.5077] | 29.33043 [27.89520 to 31.90966]
  PGT121.414.LS-D6: number analyzed (Participants) | 3 | 4 | 3 | 3 | 9 | 10
  PGT121.414.LS-D6 | 34.93493 [33.47656 to 39.49249] | 126.4765 [114.6745 to 128.2823] | 404.6015 [353.2055 to 418.2706] | 24.72877 [20.74606 to 31.10015] | 308.2920 [246.9457 to 361.4559] | 44.67182 [43.62332 to 59.62018]
  PGT121.414.LS-D84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 10
  PGT121.414.LS-D84 |  |  |  |  | 118.2193 [107.5665 to 127.2504] | 22.61336 [18.97154 to 24.21829]
  VRC07-523LS-D0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 10
  VRC07-523LS-D0 |  |  |  |  | 0.02285 [0.02285 to 0.061811] | 0.02285 [0.02285 to 0.042424]
  VRC07-523LS-D0.0417: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 8
  VRC07-523LS-D0.0417 |  |  |  |  | 630.4643 [585.8051 to 696.6382] | 0.198904 [0.131714 to 0.335898]
  VRC07-523LS-D1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 0
  VRC07-523LS-D1 |  |  |  |  | 407.5692 [365.1608 to 430.2688] |
  VRC07-523LS-D112: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 10
  VRC07-523LS-D112 |  |  |  |  | 35.65999 [27.36970 to 46.33242] | 4.320423 [3.675603 to 4.831495]
  VRC07-523LS-D112.0417: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 10
  VRC07-523LS-D112.0417 |  |  |  |  | 686.4594 [640.2608 to 810.3886] | 4.605856 [3.662888 to 5.491889]
  VRC07-523LS-D14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 10
  VRC07-523LS-D14 |  |  |  |  | 143.4822 [129.0377 to 157.1381] | 18.69117 [16.73262 to 24.82308]
  VRC07-523LS-D140: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 9
  VRC07-523LS-D140 |  |  |  |  | 122.3509 [112.0779 to 164.9094] | 21.86040 [19.27535 to 30.60428]
  VRC07-523LS-D168: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 9
  VRC07-523LS-D168 |  |  |  |  | 85.35126 [77.50010 to 86.09826] | 16.51087 [12.71702 to 18.51192]
  VRC07-523LS-D196: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 10
  VRC07-523LS-D196 |  |  |  |  | 57.95509 [42.46899 to 61.70629] | 11.16378 [9.542171 to 12.68419]
  VRC07-523LS-D224: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  VRC07-523LS-D224 |  |  |  |  | 37.81075 [26.11575 to 52.92875] | 6.780613 [6.075665 to 7.060921]
  VRC07-523LS-D224.0417: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 8
  VRC07-523LS-D224.0417 |  |  |  |  | 743.0381 [705.2543 to 786.3079] | 6.425585 [5.544769 to 8.361913]
  VRC07-523LS-D252: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 9
  VRC07-523LS-D252 |  |  |  |  | 144.2619 [34.29301 to 152.7458] | 21.76401 [19.25854 to 26.41406]
  VRC07-523LS-D28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 10
  VRC07-523LS-D28 |  |  |  |  | 102.0101 [89.62093 to 104.4785] | 15.30037 [13.04739 to 17.84672]
  VRC07-523LS-D280: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 8
  VRC07-523LS-D280 |  |  |  |  | 78.68985 [36.83790 to 92.49679] | 13.66478 [9.885758 to 17.35632]
  VRC07-523LS-D3: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 10
  VRC07-523LS-D3 |  |  |  |  | 206.2347 [203.5824 to 243.3737] | 21.27877 [18.46351 to 28.62675]
  VRC07-523LS-D336: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 9
  VRC07-523LS-D336 |  |  |  |  | 36.82022 [23.08635 to 59.66363] | 8.174529 [5.21033 to 11.59268]
  VRC07-523LS-D392: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 9
  VRC07-523LS-D392 |  |  |  |  | 18.29589 [9.388055 to 27.69066] | 4.050364 [1.956771 to 4.755294]
  VRC07-523LS-D448: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 0
  VRC07-523LS-D448 |  |  |  |  | 7.518283 [6.004015 to 15.08485] |
  VRC07-523LS-D56: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 10
  VRC07-523LS-D56 |  |  |  |  | 68.61530 [61.43403 to 78.12051] | 11.10549 [8.461712 to 11.92588]
  VRC07-523LS-D6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 10
  VRC07-523LS-D6 |  |  |  |  | 168.2826 [142.7699 to 193.8876] | 21.24964 [19.59201 to 28.91344]
  VRC07-523LS-D84: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 10
  VRC07-523LS-D84 |  |  |  |  | 49.01481 [42.62506 to 52.68755] | 7.679106 [6.178084 to 8.089730]

13. Primary Outcome: Magnitude of Serum Neutralizing Activity Measured With mAb-specific Env-pseudotyped Viruses in TZM-bl Cells
Description: Level of ID50 and ID80 titer data from the TZMbl neutralizing antibody assays against 1 bnAb-specific virus (CH505TF.N334S.N160A.N280D.1, sensitive to PGT121, resistant to VRC07) for all Part A participants (IV or SC administration of PGT121.414.LS alone), and 1 bnAb-specific virus (CNE55.N160K, sensitive to VRC07, resistant to PGT121) for all Part B participants (IV or SC administration of PGT121.414.LS in combination with VRC07523LS) at all expected timepoints.
Time Frame: Day 3, Months 1, 2, 4, 6, 8, 10, 12
Population: Overall Number of Participants Analyzed- represents the number of sampled participants. Number Analyzed shows the number of participants with available nAb data after filtering for assay specific quality control criteria at each timepoint.
Measure: Median (Inter-Quartile Range); unit: Titers
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 10 | 10
Titers
  CH505TF.N334S.N160A.N280D.1-ID50-D3: number analyzed (Participants) | 3 | 4 | 3 | 3 | 0 | 0
  CH505TF.N334S.N160A.N280D.1-ID50-D3 | 6832.5 [6821.2 to 7003.2] | 25726 [23363.6 to 28600.8] | 116600.9 [108979.7 to 133926.6] | 3427.7 [2941.7 to 4943.3] |  |
  CH505TF.N334S.N160A.N280D.1-ID50-M1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 10
  CH505TF.N334S.N160A.N280D.1-ID50-M1 |  |  |  |  | 53020.9 [28536 to 65545.7] | 5686.5 [4465.5 to 6864.9]
  CH505TF.N334S.N160A.N280D.1-ID50-M10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 8
  CH505TF.N334S.N160A.N280D.1-ID50-M10 |  |  |  |  | 32718.2 [24975.9 to 48877.2] | 5772.9 [3981.2 to 7243.8]
  CH505TF.N334S.N160A.N280D.1-ID50-M12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 9
  CH505TF.N334S.N160A.N280D.1-ID50-M12 |  |  |  |  | 39662.8 [29982.6 to 51363.2] | 6546.9 [4098 to 7237.8]
  CH505TF.N334S.N160A.N280D.1-ID50-M2 | 3890.8 [3794 to 4199.2] | 13658 [11356.2 to 16332.7] | 36244.6 [32857.4 to 70743.2] | 3448.4 [2996.3 to 5706.9] | 26629.7 [22590 to 35325.9] | 3259.5 [2769.9 to 4454.8]
  CH505TF.N334S.N160A.N280D.1-ID50-M4: number analyzed (Participants) | 3 | 4 | 3 | 3 | 9 | 10
  CH505TF.N334S.N160A.N280D.1-ID50-M4 | 2538.5 [2455.2 to 2687.3] | 5465.7 [4628.4 to 6854.7] | 18205.1 [17918.8 to 26675] | 1809 [1577 to 2057.1] | 15379 [12071.4 to 24537.5] | 2129.6 [1557.8 to 2876.5]
  CH505TF.N334S.N160A.N280D.1-ID50-M6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 9
  CH505TF.N334S.N160A.N280D.1-ID50-M6 |  |  |  |  | 46634.1 [42560.6 to 74955.6] | 7168.7 [5793.5 to 9319.8]
  CH505TF.N334S.N160A.N280D.1-ID50-M8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  CH505TF.N334S.N160A.N280D.1-ID50-M8 |  |  |  |  | 26951.7 [15555 to 42057] | 3378.6 [2734.6 to 3734.2]
  CH505TF.N334S.N160A.N280D.1-ID80-D3: number analyzed (Participants) | 3 | 4 | 3 | 3 | 0 | 0
  CH505TF.N334S.N160A.N280D.1-ID80-D3 | 2916.3 [2721.2 to 3082.5] | 9300.8 [9063.8 to 10409.4] | 45841.5 [38158.8 to 48483] | 1138 [1027.3 to 1665.6] |  |
  CH505TF.N334S.N160A.N280D.1-ID80-M1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 10
  CH505TF.N334S.N160A.N280D.1-ID80-M1 |  |  |  |  | 17845.1 [10766.7 to 23337] | 1905.1 [1624.7 to 2328]
  CH505TF.N334S.N160A.N280D.1-ID80-M10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 8
  CH505TF.N334S.N160A.N280D.1-ID80-M10 |  |  |  |  | 13884.8 [7506.2 to 15979.8] | 1658.2 [1217.5 to 2494.5]
  CH505TF.N334S.N160A.N280D.1-ID80-M12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 9
  CH505TF.N334S.N160A.N280D.1-ID80-M12 |  |  |  |  | 12040.2 [7037.7 to 14895.8] | 1366.9 [958.9 to 1765.3]
  CH505TF.N334S.N160A.N280D.1-ID80-M2 | 1320.9 [1313.7 to 1402.3] | 4458.1 [3360.6 to 5606.9] | 12014.8 [11496.4 to 23690.5] | 1238.9 [1220 to 1736.6] | 9708.8 [7510.3 to 13896.2] | 1150.6 [962.4 to 1620.9]
  CH505TF.N334S.N160A.N280D.1-ID80-M4: number analyzed (Participants) | 3 | 4 | 3 | 3 | 9 | 10
  CH505TF.N334S.N160A.N280D.1-ID80-M4 | 712.2 [688.9 to 739] | 2144.3 [1727.6 to 2608.7] | 6949.7 [6162.4 to 8432.2] | 573.6 [561.5 to 727.9] | 4439.9 [3907.5 to 6936.3] | 555.2 [506.1 to 675.3]
  CH505TF.N334S.N160A.N280D.1-ID80-M6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 9
  CH505TF.N334S.N160A.N280D.1-ID80-M6 |  |  |  |  | 17924.3 [16013.6 to 18093.5] | 1803.7 [1688.6 to 2319.2]
  CH505TF.N334S.N160A.N280D.1-ID80-M8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  CH505TF.N334S.N160A.N280D.1-ID80-M8 |  |  |  |  | 6137.5 [5157.2 to 12462.7] | 1074.3 [936 to 1347.5]
  CNE55.N160K-ID50-M1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 10
  CNE55.N160K-ID50-M1 |  |  |  |  | 1644.8 [889.9 to 2377.7] | 50.4 [34.1 to 80.9]
  CNE55.N160K-ID50-M10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 8
  CNE55.N160K-ID50-M10 |  |  |  |  | 881.4 [296.7 to 2596.9] | 67 [35 to 103.7]
  CNE55.N160K-ID50-M12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 9
  CNE55.N160K-ID50-M12 |  |  |  |  | 394.1 [139 to 730.3] | 57.5 [23.1 to 82.4]
  CNE55.N160K-ID50-M2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 10
  CNE55.N160K-ID50-M2 |  |  |  |  | 1197.6 [564.5 to 2642.1] | 45.9 [33.2 to 56.7]
  CNE55.N160K-ID50-M4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 10
  CNE55.N160K-ID50-M4 |  |  |  |  | 183.5 [110.7 to 669] | 5 [5 to 5]
  CNE55.N160K-ID50-M6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 9
  CNE55.N160K-ID50-M6 |  |  |  |  | 1088 [508.5 to 3589.4] | 66.2 [39.2 to 69]
  CNE55.N160K-ID50-M8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  CNE55.N160K-ID50-M8 |  |  |  |  | 318.2 [118.9 to 765.2] | 15.8 [5 to 28.9]
  CNE55.N160K-ID80-M1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 10
  CNE55.N160K-ID80-M1 |  |  |  |  | 258.6 [135.5 to 312.8] | 5 [5 to 5]
  CNE55.N160K-ID80-M10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 8
  CNE55.N160K-ID80-M10 |  |  |  |  | 151.9 [32.1 to 183.7] | 5 [5 to 5]
  CNE55.N160K-ID80-M12: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 9
  CNE55.N160K-ID80-M12 |  |  |  |  | 34.9 [26.9 to 73.4] | 5 [5 to 5]
  CNE55.N160K-ID80-M2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 10
  CNE55.N160K-ID80-M2 |  |  |  |  | 111.9 [65.9 to 201.6] | 7.6 [5 to 12.1]
  CNE55.N160K-ID80-M4: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 10
  CNE55.N160K-ID80-M4 |  |  |  |  | 37.4 [32.2 to 68.6] | 5 [5 to 5]
  CNE55.N160K-ID80-M6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 9
  CNE55.N160K-ID80-M6 |  |  |  |  | 130.5 [105.1 to 198.4] | 5 [5 to 14]
  CNE55.N160K-ID80-M8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  CNE55.N160K-ID80-M8 |  |  |  |  | 29 [20.6 to 41.5] | 5 [5 to 5]

14. Secondary Outcome: Occurrence of Antidrug Antibodies (ADA)
Description: Antidrug antibodies (ADA) are most typically detected and characterized using a tiered testing strategy. In Tier I, a sensitive binding assay is used to determine if samples may have ADA present. In Tier II, the response is confirmed, typically by establishing the specificity of the response by competition with free drug. In Tier III, the response is characterized, typically with a neutralization reduction assay and/or a titering assay.
Time Frame: Day 0, 112, 196, 224, 336, 392, 448
Population: Overall Number of Participants Analyzed presents the number of enrolled participants in each treatment arm. Number Analyzed shows the number of samples available and tested in a certain tier and timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 10 | 10
Participants
  PGT121.414.LS-Tier I-D0 | 0 | 0 | 0 | 0 | 0 | 0
  PGT121.414.LS-Tier I-D112: number analyzed (Participants) | 3 | 4 | 3 | 3 | 9 | 10
  PGT121.414.LS-Tier I-D112 | 0 | 0 | 0 | 0 | 0 | 0
  PGT121.414.LS-Tier I-D196: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 10
  PGT121.414.LS-Tier I-D196 |  |  |  |  | 0 | 0
  PGT121.414.LS-Tier I-D224: number analyzed (Participants) | 3 | 4 | 3 | 0 | 9 | 9
  PGT121.414.LS-Tier I-D224 | 0 | 0 | 0 |  | 0 | 0
  PGT121.414.LS-Tier I-D336: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 9
  PGT121.414.LS-Tier I-D336 |  |  |  |  | 0 | 0
  PGT121.414.LS-Tier I-D392: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 9
  PGT121.414.LS-Tier I-D392 |  |  |  |  | 0 | 0
  PGT121.414.LS-Tier I-D448: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 0
  PGT121.414.LS-Tier I-D448 |  |  |  |  | 0 |
  VRC07-523LS-Tier I-D0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 10 | 10
  VRC07-523LS-Tier I-D0 |  |  |  |  | 1 | 0
  VRC07-523LS-Tier I-D112: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 10
  VRC07-523LS-Tier I-D112 |  |  |  |  | 0 | 0
  VRC07-523LS-Tier I-D196: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 10
  VRC07-523LS-Tier I-D196 |  |  |  |  | 0 | 0
  VRC07-523LS-Tier I-D224: number analyzed (Participants) | 0 | 0 | 0 | 0 | 9 | 9
  VRC07-523LS-Tier I-D224 |  |  |  |  | 0 | 0
  VRC07-523LS-Tier I-D336: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 9
  VRC07-523LS-Tier I-D336 |  |  |  |  | 0 | 0
  VRC07-523LS-Tier I-D392: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 9
  VRC07-523LS-Tier I-D392 |  |  |  |  | 0 | 0
  VRC07-523LS-Tier I-D448: number analyzed (Participants) | 0 | 0 | 0 | 0 | 7 | 0
  VRC07-523LS-Tier I-D448 |  |  |  |  | 0 |
  VRC07-523LS-Tier II-D0: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 0
  VRC07-523LS-Tier II-D0 |  |  |  |  | 0 |

15. Secondary Outcome: Magnitude and Breadth of Neutralizing Antibody Responses Against Autologous Viral Isolates as Assessed by Area Under the Magnitude-breadth Curves at Months 1, 4, and 9
Description: Magnitude-breadth characterize the magnitude (ID50 or ID80 titers) and breadth (number of virus isolates) of each individual serum sample assayed against a panel of virus isolates. MB curves show, for each possible magnitude threshold, the fraction of assays with magnitudes greater than this threshold. The area under the magnitude-breadth curve (AUC-MB) is calculated as the average of the log10-based ID50 or ID80 titers over the panel of isolates. Isolates includes: 0330.v4.c3, 3426.v5.c17, 377.v4.c09, AC10.0.29, Ce1176_A3, DU156.12, DU172.17, PVO.4, RHPA4259.7, SC422661.8, T2638, andTRO.11.
Time Frame: Months 1, 4, and 9
Population: as for outcome 14
Measure: Median (Inter-Quartile Range); unit: log10(titer)
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine
Number analyzed (Participants) | 3 | 4 | 3 | 3 | 10 | 10
log10(titer)
  ID50-M1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 9 | 7
  ID50-M1 | 2.87 [2.86 to 2.99] | 3.39 [3.38 to 3.42] | 4 [3.91 to 4.14] | 2.79 [2.78 to 2.89] | 3.97 [3.92 to 4.01] | 3.02 [2.97 to 3.07]
  ID50-M4: number analyzed (Participants) | 3 | 4 | 3 | 3 | 0 | 0
  ID50-M4 | 2.54 [2.5 to 2.57] | 3.08 [2.99 to 3.15] | 3.55 [3.44 to 3.58] | 2.42 [2.39 to 2.61] |  |
  ID50-M9: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 7
  ID50-M9 |  |  |  |  | 4.12 [3.65 to 4.22] | 3.2 [3.17 to 3.27]
  ID80-M1: number analyzed (Participants) | 3 | 3 | 3 | 3 | 9 | 7
  ID80-M1 | 2.28 [2.28 to 2.36] | 2.84 [2.83 to 2.84] | 3.36 [3.29 to 3.48] | 2.23 [2.15 to 2.29] | 3.46 [3.4 to 3.49] | 2.47 [2.44 to 2.51]
  ID80-M4: number analyzed (Participants) | 3 | 4 | 3 | 3 | 0 | 0
  ID80-M4 | 1.89 [1.85 to 1.91] | 2.36 [2.24 to 2.49] | 2.88 [2.82 to 2.97] | 1.81 [1.79 to 1.92] |  |
  ID80-M9: number analyzed (Participants) | 0 | 0 | 0 | 0 | 8 | 7
  ID80-M9 |  |  |  |  | 3.62 [3.06 to 3.71] | 2.66 [2.65 to 2.71]

ADVERSE EVENTS:
Time Frame: Measured through Month 24 for Unsolicited AEs and Measured through 3 days after each vaccine dose at T1-T4: Day 0; T5-T6: Days 0, 112, 224 for Solicited AEs
Description: The number (percentage) of Participants Reporting Solicited AEs and unsolicited AEs including All-Cause Mortality, Serious Adverse Events (SAEs), and Other (Not Including Serious) Adverse Events ware summarized by arm
Arm/Group | Group 1: Vaccine | Group 2: Vaccine | Group 3: Vaccine | Group 4: Vaccine | Group 5: Vaccine | Group 6: Vaccine
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 2/3 | 10/10 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Vaccine (N=3) | Group 2: Vaccine (N=3) | Group 3: Vaccine (N=3) | Group 4: Vaccine (N=3) | Group 5: Vaccine (N=10) | Group 6: Vaccine (N=10)
Bundle branch block left (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Solicited) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (Solicited) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Infusion site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site erythema (Solicited) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Infusion site pain (Solicited) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 7 (7)
Infusion site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site swelling (Solicited) (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Malaise (Solicited) (General disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 6 (6) | 5 (5)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Dermatophytosis of nail (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 1 (1)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body temperature increased (Solicited) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Solicited) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Solicited) (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (Solicited) (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 7 (7) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Premenstrual dysphoric disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Solicited) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria cholinergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-10-08): https://cdn.clinicaltrials.gov/large-docs/91/NCT04212091/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/91/NCT04212091/SAP_001.pdf